CLINICAL TRIAL: NCT06965387
Title: Deep Learning-Based Evaluation of Gummy Smile: Development and Validation of a Segmentation Model
Brief Title: Deep Learning for Gummy Smile Segmentation
Status: Recruiting | Type: Observational
Sponsor: Gazi University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Gülenay Çolak, Research Assistant, Gazi University
Other Study IDs: E-77082166-604.01-881629
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Gummy Smile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- • High smile: Gingival margins and cervical areas are clearly visible above the upper lip line.

SUMMARY:
A gummy smile (excessive visibility of the gums when smiling) is not merely an aesthetic issue but also an important parameter in terms of periodontal health. Current evaluation methods are subjective and non-standardized, leading to limitations in both clinical accuracy and patient communication. In recent years, AI-based models have begun to be effectively used in dental image analysis and diagnostic processes. This study aims to develop an AI-supported objective and reproducible analysis model capable of evaluating gummy smile from both aesthetic and periodontal perspectives using a unique dataset composed of images obtained through standard clinical protocols and labeled by the same expert.

Individuals aged 12 years or older with no maxillary anterior (teeth #13-23) tooth loss will be included in the study. Patients with missing anterior maxillary teeth (teeth #13-23), significant anatomical pathologies, or smile-interfering factors (e.g., facial piercings, orthodontic appliances, facial hair) will be excluded.

Standardized frontal photographs will be taken using a single device (iPhone 15) to ensure consistency in resolution, lighting, and color balance. Images will be captured from a fixed distance of 15 cm with participants in an upright position, eyes facing forward, and heads aligned to the Frankfurt Horizontal Plane. To maintain standardization, the smartphone's grid lines will be used to align the horizontal line with the pupils and vertical lines with the nasal alae.

Images of high, average, and low smile lines will be labeled by a periodontist using the web-based annotation tool MakeSense. Visible gingival areas will be annotated as polygons bounded superiorly by the lower border of the upper lip and inferiorly by the gingival margin. For participants with high smile lines, gingival display will be measured using ImageJ (National Institutes of Health, Bethesda, MD, USA), with calibration performed via a periodontal probe embedded in each photo. A pixel-to-millimeter conversion factor will be derived and applied to measurements between the upper lip and gingival margin in the anterior maxillary sextant (teeth #13-23). Distances between paired landmarks (points 7-13, 8-14, 9-15, 10-16, 11-17, 12-18) will be measured in millimeters. AI-based segmentation outputs (via MakeSense) will be statistically compared to ImageJ measurements to assess correlation.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 12 years or older with no maxillary anterior (teeth #13-23) tooth loss will be included in the study.

Exclusion Criteria:

* Patients with missing anterior maxillary teeth (teeth #13-23), significant anatomical pathologies, or smile-interfering factors (e.g., facial piercings, orthodontic appliances, facial hair) will be excluded.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who presented to the Department of Periodontology, Faculty of Dentistry, Gazi University, for routine dental evaluation and treatment
Sampling Method: Non-Probability Sample
Enrollment: 1740 (Estimated)
Dates: Start 2025-01-12 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Evaluation of gummy samples using artificial intelligence | From enrollment to the end of treatment at 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Turgut Cankaya, Associate Professor, Study Director — Gazi University
Locations (1):
- Gazi University, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided